CLINICAL TRIAL: NCT06609382
Title: Prognostic Value of Left Ventricular Mass Index in Obstructive Hypertrophic Cardiomyopathy Undergoing Septal Myectomy
Brief Title: Left Ventricular Mass Index Predicts Clinical Outcomes in Patients with Obstructive Hypertrophic Cardiomyopathy Undergoing Septal Myectomy
Acronym: LVMI and oHCM
Status: Completed | Type: Observational
Sponsor: Changrong Nie (Other)
Responsible Party: Sponsor-Investigator, Changrong Nie, MD, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Other Study IDs: 2020-1315; 2022-GSP-GG-29 (Other Grant/Funding Number: National High Level Hospital Clinical Research Funding)
Record Dates: First submitted 2024-09-21; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy (oHCM)
Keywords: left ventricular mass index; all-cause death; survival; obstructive hypertrophic cardiomyopathy; septal myectomy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Obstructive hypertrophic cardiomyopathy who underwent septal myectomy: Patients who had at least one cardiac magnetic resonance examination before surgery.
  Interventions: Other: Patients had a higher left ventricular mass index or not （the exact value is determined by the cut-off value for the clinical outcomes)

INTERVENTIONS:
Other: Patients had a higher left ventricular mass index or not （the exact value is determined by the cut-off value for the clinical outcomes) — Patients were grouped by the cutoff value of left ventricular mass index (LVMI) for all cause death, and the Maximally Selected Rank Statistics method was used to determine the optimal cutoff point of LVMI for death.

SUMMARY:
In this study, we aimed to analyze the association between left ventricular mass index and clinical outcomes to provide the potential indicator for worse survival.

DETAILED DESCRIPTION:
This retrospective study aimed to determine the prognostic value of left ventricular mass index in predicting clinical outcomes, including all-cause death, new-onset or recurrent atrial fibrillation, and a composite endpoint of all-cause death, heart failure,permanent pacemaker implantation, new-onset or recurrent atrial fibrillation, and stroke.

ELIGIBILITY:
Inclusion Criteria:(1) Difficulty in relieving symptoms with medication or recurrent syncope. (2) Left ventricular outflow tract (LVOT) pressure gradient ≥ 50 mmHg at rest or with provocation and the maximum thickness of the septum is ≧ 15 mm.

Exclusion Criteria:

* (1) Combined right ventricular outflow tract obstruction requiring right ventricular outflow tract dissection. (2) Combined mitral or aortic valve organic lesions requiring valve replacement surgery. (3) Apical ventricular aneurysm formation requiring ventriculotomy. (4) Previous septal reduction therapy, including alcohol ablation or septal myectomy. (5) patients did not undergo cardiac magnetic resonance examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: oHCM who underwent septal myectomy and had at least one CMR image before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause death | One month after discharge
  Any death observed one month after discharge.

SECONDARY OUTCOMES:
composite endpoint | One month after discharge
  Composite endpoint included all-cause death, and nonfatal adverse events, with nonfatal adverse events defined as rehospitalization for heart failure, permanent pacemaker implantation, new-onset or recurrent atrial fibrillation, and stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No